CLINICAL TRIAL: NCT06313047
Title: Pharmacogenetic of Doxorubicin in Patients With Hepatocellular Carcinoma: A Prospective Cohort Study
Brief Title: Pharmacogenetic of Doxorubicin in HCC.
Status: Completed | Type: Observational
Sponsor: Rehab Werida (Other)
Collaborators: King Saud Bin Abdulaziz University for Health Sciences (Other); King Abdulaziz University (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Associate Professor, Damanhour University
Organization: Damanhour University (Other)
Other Study IDs: Doxorubacin in HCC
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC patients: Each of the patients was given Doxorubicin and followed up for one year.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — each recruited patient with HCC received a comprehensive review of their medical history, physical status, and laboratory results.
  Other Names: Dox

SUMMARY:
The study included 81 HCC patients, both male and female. Prior to being assessed for eligibility, each recruited patient with HCC received a comprehensive review of their medical history, physical status, and laboratory results. Every research participant take part in the experiment and provided written informed consent.

DETAILED DESCRIPTION:
All patients had their baseline viral indicators for HBV and HCV evaluated. Additionally, blood samples were taken for genotyping. All patients underwent evaluations of their kidney, liver, and alpha fetoprotein (AFP) functions, as well as their complete blood count (CBC), at both the baseline and follow-up appointments. To evaluate the efficacy of TACE, triple pelvic abdominal CT scans were performed both prior to and one month later. Using triphasic pelviabdominal CT, patients who achieved complete response (CR) were monitored for up to 13 months following chemotherapy in order to identify recurrence. Follow-up appointments were planned to identify patients responces or any negative effects.

ELIGIBILITY:
Inclusion Criteria:

1. When diagnosing the patient with HCC, the guidelines provided by the American Association for the Study of Liver Diseases (AASLD) were adhered to.
2. Be above 20 years old.
3. Individuals with intact organs.
4. There is no cure for HCC in surgery, microwave treatment, or radiofrequency ablation.

Exclusion Criteria:

1. The patients refused to sign the formal consent.
2. Be more than 75 years old.
3. There is a notable case of portal vein thrombosis.
4. Spreads beyond the liver.
5. Encephalopathy of the liver.
6. Present sickness.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 HCC patients, both male and female. Prior to being assessed for eligibility, each recruited patient with HCC received a comprehensive review of their medical history, physical status, and laboratory results.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
GSTP1 | 1 year
  Genotyping
CYP2B6 | 1 year
  Genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Sireen Shilbayeh, Prof., Study Chair — Princess Nourah Bint Abdul Rahman University; Mohammad A. Alshabeeb, Study Director — King Saud Bin Abdulaziz University for Health Sciences; Abdalrhman H Alanizi, Principal Investigator — King Abdulaziz University; Naglaa Khedr, Prof., Study Director — Tanta University
Locations (1):
- King Abdullah bin Abdulaziz University Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Shilbayeh SAR, Abd El-Baset OA, Alshabeeb MA, Alanizi AH, Khedr NF, Werida RH. The Influence of CYP2B6, GSTP1, and SLCO1B1 Star Allele-Predicted Phenotypes and CBR1 Genetic Variants on Effectiveness Outcomes in Patients With Hepatocellular Carcinoma Receiving Doxorubicin via Transarterial Chemoembolization. Pharmacol Res Perspect. 2025 Jun;13(3):e70114. doi: 10.1002/prp2.70114. PMID 40405401